CLINICAL TRIAL: NCT03872453
Title: Phase II/III: Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Trial of BHV-3500 for the Acute Treatment of Migraine
Brief Title: Acute Treatment Trial in Adult Subjects With Migraines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3500-201
Record Dates: First submitted 2019-03-06; First posted 2019-03-13 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Migraine
Keywords: Acute Migraine; phonophobia; photophobia; nausea
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Subject
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Zavegepant 5 mg (Experimental): Participants administered a single intranasal dose of zavegepant 5 mg on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar Unidose System (UDS) liquid spray device.
  Interventions: Drug: Zavegepant; Device: Intranasal Aptar Pharma Unit Dose System
- Zavegepant 10 mg (Experimental): Participants administered a single intranasal dose of zavegepant 10 mg on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar UDS liquid spray device.
  Interventions: Drug: Zavegepant; Device: Intranasal Aptar Pharma Unit Dose System
- Zavegepant 20 mg (Experimental): Participants administered a single intranasal dose of zavegepant 20 mg on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar UDS liquid spray device.
  Interventions: Drug: Zavegepant; Device: Intranasal Aptar Pharma Unit Dose System
- Placebo (Placebo Comparator): Participants administered a single intranasal dose of zavegepant-matching placebo on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar UDS liquid spray device.
  Interventions: Drug: Zavegepant matching placebo; Device: Intranasal Aptar Pharma Unit Dose System

INTERVENTIONS:
Drug: Zavegepant — A single dose of zavegepant
  Other Names: BHV3500
  Arms: Zavegepant 10 mg; Zavegepant 20 mg; Zavegepant 5 mg
Drug: Zavegepant matching placebo — A single dose of placebo matched to zavegepant
  Arms: Placebo
Device: Intranasal Aptar Pharma Unit Dose System — A single-dose intranasal device

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of three different intranasal dose levels of zavegepant (BHV-3500), relative to placebo, in the acute treatment of moderate to severe migraine.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Participants have at least 1-year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, including the following:

1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age.
2. Migraine attacks, on average, lasting about 4-72 hours if untreated.
3. Not more than 8 attacks of moderate to severe intensity per month within the last 3 months.
4. At least 2 consistent migraine headache attacks of moderate or severe intensity in each of the 3 months prior to the Screening Visit and throughout the Screening Period.
5. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to the Screening Visit and throughout the Screening Period.
6. Participants on prophylactic migraine medication are permitted to remain on therapy provided they have been on a stable dose for at least 3 months prior to Screening Visit and the dose is not expected to change during the course of the study.
7. Participants with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Exclusion Criteria:

Key Exclusion Criteria:

1. Participant with a history of basilar migraine or hemiplegic migraine.
2. Participant with a history of human immunodeficiency virus (HIV) disease.
3. Participant history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Participants with myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, cardiac surgery, stroke or transient ischemic attack during the 6 months prior to screening.
4. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to being enrolled).
5. Participant has a current diagnosis of major depression, other pain syndromes, psychiatric conditions (for example, schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion might interfere with study assessments.
6. Participant has a history of gastric, or small intestinal surgery (including gastric bypass, gastric banding, gastric sleeve, gastric balloon, etc.), or has disease that causes malabsorption.
7. The participant has a history of current or evidence of any significant and/ or unstable medical conditions (for example, history of congenital heart disease or arrhythmia, known suspected infection, hepatitis B or C, or cancer) that, in the Investigator's opinion, would expose them to undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial.
8. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or subjects who have met Diagnostic and Statistical Manual of Mental Disorders Fifth edition (DSM-V) criteria for any significant substance use disorder within the past 12 months from the date of the Screening Visit.
9. History of nasal surgery in the 6 months preceding the Screening Visit.
10. Participation in any other investigational clinical trial while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2154 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (82):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Pharmacology Research Institute, Encino, California
  - eStudySite, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - National Research Institute, Panorama City, California
  - Optimus Medical Group, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Denver Neurological Research, LLC, Denver, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Ki Health Partners, LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - MD Clinical, Hallandale, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - AGA Clinical Trials, Miami, Florida
  - Qps Mra, Llc, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Meridien Research, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Family Medicine Specialists/CIS, Wauconda, Illinois
  - Phoenix Medical Research, Prairie Village, Kansas
  - Crescent City Headache and Neurology Center, LLC, Chalmette, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Community Clinical Research Network, Marlborough, Massachusetts
  - Regeneris Medical, North Attleboro, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - Clinical Research Institute, Inc., Plymouth, Minnesota
  - MedPharmics, LLC, Biloxi, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Meritas Health Neurology, North Kansas City, Missouri
  - QPS Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Montefiore Medical Center: Headache Center, The Bronx, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Alliance for Multispecialty Research/New Orleans Center for Clinical Research/Volunteer Research, Knoxville, Tennessee
  - Clinical Neuroscience Solutions DBA CNS Healthcare, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Star Research, LLC, Lake Jackson, Texas
  - Advanced Pharmaceutical Development Clinical Research, Magnolia, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Dynamed Clinical Research, Tomball, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research, Bellevue, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3500-201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 82 sites in the United States.
Pre-assignment Details: A total of 2154 participants were enrolled, of which 1673 participants were randomized in a 1:1:1:1 ratio across the 4 treatment groups into the zavegepant (5 mg, 10 mg, or 20 mg) or placebo treatment groups. The randomization was stratified by the use of prophylactic migraine medications (yes or no). 481 participants were not randomized due to lost to follow-up, screen failure, withdrawal by participants, or other reasons.
Period: Overall Study
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Started (Randomized) | 418 | 417 | 418 | 420
Treated | 388 | 394 | 403 | 403
Modified Intent-to-Treat (mITT) Participants (Treated participants who were randomized only once, had moderate to severe pain at on-study migraine attack onset, and had non-missing, post-baseline efficacy data.) | 387 | 391 | 402 | 401
Completed | 386 | 391 | 399 | 402
Not Completed | 32 | 26 | 19 | 18
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 8 | 7 | 4 | 4
Not completed — Never Treated Migraine | 19 | 17 | 13 | 12
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Other Than Specified | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Participants included enrolled participants who took study therapy (zavegepant or placebo).
Groups:
- Zavegepant 5 mg: Participants administered a single intranasal dose of zavegepant 5 mg on occurrence of migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar UDS liquid spray device.
- Zavegepant 20 mg: Participants administered a single intranasal dose of zavegepant 20 mg migraine that reached moderate or severe intensity within 45 days after randomization. The dose was administered using Aptar UDS liquid spray device.
- Total: Total of all reporting groups
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo | Total
Number analyzed (Participants) | 388 | 394 | 403 | 403 | 1588
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (12.58) | 41.3 (12.96) | 40.0 (12.95) | 40.0 (12.07) | 40.8 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337 | 335 | 344 | 338 | 1354
  Male | 51 | 59 | 59 | 65 | 234
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 69 | 72 | 81 | 286
  Not Hispanic or Latino | 324 | 325 | 331 | 322 | 1302
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 3 | 1 | 6
  Asian | 17 | 13 | 15 | 13 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 65 | 74 | 62 | 59 | 260
  White | 299 | 297 | 316 | 329 | 1241
  More than one race | 5 | 9 | 7 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Prophylactic migraine medication use at randomization [Count of Participants; unit: Participants]
  Yes | 54 | 50 | 57 | 55 | 216
  No | 334 | 344 | 346 | 348 | 1372

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Pain at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the electronic clinical outcome assessment (eCOA) handheld device. Pain freedom was defined as pain level of none post-dose.
Time Frame: 2 hours post-dose
Population: mITT participants included treated participants who were randomized only once, had moderate to severe pain at on-study migraine attack onset, and had non-missing, post-baseline efficacy data.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 19.6 [14.8 to 24.5] | 22.5 [17.5 to 27.6] | 23.1 [18.1 to 28.2] | 15.5 [11.1 to 19.8]
Statistical Analysis 1: Comparison: Zavegepant 5 mg vs Placebo; Test type: Superiority — The stratified percentage difference between zavegepant group and placebo was tested at a Bonferroni-corrected alpha level of 0.0167; p = 0.1214, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 4.2, 98.3% CI 2-sided [-2.3 to 10.7]
Statistical Analysis 2: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0113, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 7.0, 98.3% CI 2-sided [0.4 to 13.7]
Statistical Analysis 3: Comparison: Zavegepant 20 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0055, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 7.7, 98.3% CI 2-sided [1.1 to 14.3]

2. Primary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-dose
Description: MBS was reported as nausea, photophobia, or phonophobia at migraine onset using the eCOA handheld device. Symptom status (absent, present) was assessed post-dose using the eCOA handheld device separately for nausea, photophobia, and phonophobia. Freedom from MBS was defined as MBS reported at on-study migraine attack onset that was absent post-dose.
Time Frame: 2 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 39.0 [33.1 to 45.0] | 41.9 [36.0 to 47.9] | 42.5 [36.6 to 48.4] | 33.7 [28.0 to 39.3]
Statistical Analysis 1: Comparison: Zavegepant 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1162, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 5.4, 98.3% CI 2-sided [-2.8 to 13.6]
Statistical Analysis 2: Comparison: Zavegepant 10 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0155, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 8.3, 98.3% CI 2-sided [0.1 to 16.5]
Statistical Analysis 3: Comparison: Zavegepant 20 mg vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0094, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 8.9, 98.3% CI 2-sided [0.7 to 17.0]

3. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Pain relief was defined as pain level of none or mild.
Time Frame: 2 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 57.9 [51.9 to 63.9] | 60.6 [54.7 to 66.5] | 61.2 [55.4 to 67.0] | 53.6 [47.7 to 59.6]
Statistical Analysis 1: Comparison: Zavegepant 10 mg vs Placebo; If the coprimary endpoint tests were both significant for a zavegepant dose group versus placebo, the secondary endpoints were tested for that zavegepant dose group versus placebo using a hierarchical gate-keeping procedure in the order the endpoints are reported, with each test in the hierarchy conducted at alpha = 0.0167. If a test in the hierarchy was not significant, any further tests on endpoints in the sequence were not considered significant for any zavegepant dose group versus placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0439, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 7.1, 98.3% CI 2-sided [-1.3 to 15.4]
Statistical Analysis 2: Comparison: Zavegepant 20 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0302, Cochran-Mantel-Haenszel — Threshold for significance at 0.0167 level; Stratified Percentage Difference = 7.5, 98.3% CI 2-sided [-0.8 to 15.9]

4. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 2 Hours Post-dose
Description: Functional disbaility level was assessed on a 4-point scale (normal function, mildly impaired, severely impaired, requires bedrest) using the eCOA handheld device. Normal function was defined as a functional disability level of normal post-dose in the subset of participants with functional disability (mildly impaired, severely impaired, requires bedrest) at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The mITT participants with functional disability at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 363 | 354 | 372 | 369
percentage of participants | 31.7 [25.8 to 37.5] | 34.5 [28.4 to 40.5] | 34.7 [28.8 to 40.6] | 27.4 [21.8 to 32.9]

5. Secondary Outcome: Percentage of Participants With Rescue Medication Use Within 24 Hours Post-dose
Description: Participants who did not experience relief of their migraine headache at the end of 2 hours after dosing with study medication (and after the 2-hour assessments had been completed on the eCOA handheld device) were permitted to use the following rescue medications: aspirin, ibuprofen, acetaminophen up to 1000 mg/day (this includes Excedrin® Migraine), naproxen (or any other type of nonsteroidal anti-inflammatory drug), antiemetics (for example, metoclopramide or promethazine), or baclofen. The participant's use of rescue medication was recorded by the site on a case report form.
Time Frame: Through 24 hours post-dose
Population: The mITT participants were analyzed. Participants with rescue medication start date less than or equal to (≤) study drug start date + 1 day and missing rescue medication start time were excluded.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 385 | 388 | 397 | 400
percentage of participants | 24.9 [19.7 to 30.2] | 26.0 [20.7 to 31.4] | 20.2 [15.3 to 25.0] | 27.3 [21.9 to 32.6]

6. Secondary Outcome: Percentage of Participants With Freedom From Photophobia at 2 Hours Post-dose
Description: Photophobia (sensitivity to light) status was measured as absent or present in the eCOA handheld device. Freedom from photophobia was defined as photophobia absent post-dose in the subset of participants with photophobia present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The mITT participants with symptom of photophobia present at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 337 | 340 | 354 | 358
percentage of participants | 35.0 [28.8 to 41.2] | 35.6 [29.4 to 41.8] | 37.9 [31.7 to 44.0] | 30.4 [24.6 to 36.3]

7. Secondary Outcome: Percentage of Participants With Freedom From Phonophobia at 2 Hours Post-dose
Description: Phonophobia (sensitivity to sound) status was measured as absent or present in the eCOA handheld device. Freedom from phonophobia was defined as phonophobia absent post-dose in the subset of participants with phonophobia present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The mITT participants with symptom of phonophobia present at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 260 | 239 | 263 | 276
percentage of participants | 44.2 [36.9 to 51.6] | 44.8 [37.1 to 52.5] | 43.3 [36.0 to 50.7] | 34.1 [27.2 to 40.9]

8. Secondary Outcome: Percentage of Participants With Pain Relief at 60 Minutes Post-dose
Description: as for outcome 3
Time Frame: 60 minutes post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 47.0 [41.0 to 53.1] | 46.0 [40.0 to 52.1] | 49.8 [43.8 to 55.7] | 41.9 [36.0 to 47.8]

9. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 60 Minutes Post-dose
Description: as for outcome 4
Time Frame: 60 minutes post-dose
Population: The mITT participants with functional disability at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 363 | 354 | 372 | 369
percentage of participants | 22.6 [17.3 to 27.8] | 18.9 [13.9 to 23.9] | 18.8 [14.0 to 23.7] | 17.1 [12.4 to 21.8]

10. Secondary Outcome: Percentage of Participants With Pain Relief at 30 Minutes Post-dose
Description: as for outcome 3
Time Frame: 30 minutes post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 26.6 [21.2 to 32.0] | 29.9 [24.4 to 35.5] | 26.6 [21.3 to 31.9] | 24.7 [19.5 to 29.8]

11. Secondary Outcome: Percentage of Participants Who Were Able to Function Normally at 30 Minutes Post-dose
Description: as for outcome 4
Time Frame: 30 minutes post-dose
Population: The mITT participants with functional disability at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 363 | 354 | 372 | 369
percentage of participants | 8.8 [5.3 to 12.4] | 7.6 [4.2 to 11.0] | 9.9 [6.2 to 13.7] | 5.4 [2.6 to 8.2]

12. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 43.7 [37.6 to 49.7] | 42.5 [36.5 to 48.4] | 44.5 [38.6 to 50.5] | 35.7 [29.9 to 41.4]

13. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain freedom was defined as pain level of none at 2 hours up to 24 hours post-dose.
Time Frame: From 2 hours up to 24 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 14.2 [10.0 to 18.5] | 15.1 [10.8 to 19.4] | 15.7 [11.3 to 20.0] | 9.0 [5.6 to 12.4]

14. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain relief was defined as pain level of none or mild at 2 hours up to 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 40.1 [34.1 to 46.0] | 39.6 [33.7 to 45.6] | 38.8 [33.0 to 44.6] | 32.7 [27.1 to 38.3]

15. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Sustained pain freedom was defined as pain level of none at 2 hours up to 48 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The mITT participants were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 387 | 391 | 402 | 401
percentage of participants | 12.9 [8.8 to 17.0] | 13.8 [9.6 to 18.0] | 13.2 [9.1 to 17.2] | 7.5 [4.3 to 10.6]

16. Secondary Outcome: Percentage of Participants With Freedom From Nausea at 2 Hours Post-dose
Description: Nausea status was measured as absent or present in the eCOA handheld device. Freedom from nausea was defined as nausea absent post-odse in the subset of participants with nausea present at on-study migraine attack onset.
Time Frame: 2 hours post-dose
Population: The mITT participants with symptom of nausea present at on-study migraine attack onset were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 237 | 243 | 265 | 239
percentage of participants | 53.2 [45.4 to 60.9] | 53.9 [46.3 to 61.6] | 54.7 [47.4 to 62.0] | 51.0 [43.3 to 58.8]

17. Secondary Outcome: Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-dose
Description: Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eCOA handheld device. Pain relapse was defined as pain level of mild, moderate, or severe after 2 hours up to 48 hours post-dose in the subset of participants with pain level of none at 2 hours post-dose.
Time Frame: From 2 hours up to 48 hours post-dose
Population: The mITT participants with pain freedom at 2 hours post-dose were analyzed.
Measure: Number (98.3% Confidence Interval); unit: percentage of participants
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
Number analyzed (Participants) | 76 | 88 | 93 | 62
percentage of participants | 31.6 [18.8 to 44.3] | 33.0 [21.0 to 45.0] | 37.6 [25.6 to 49.7] | 50.0 [34.8 to 65.2]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from study drug dosing up to the end of the study (up to 52 days).
Description: Treated Participants included enrolled participants who took study therapy (zavegepant or placebo).
Arm/Group | Zavegepant 5 mg | Zavegepant 10 mg | Zavegepant 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/388 | 0/394 | 0/403 | 0/403
Serious Adverse Events (participants affected / at risk) | 0/388 | 1/394 | 0/403 | 1/403
Other Adverse Events (participants affected / at risk) | 57/388 | 58/394 | 81/403 | 15/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 5 mg (N=388) | Zavegepant 10 mg (N=394) | Zavegepant 20 mg (N=403) | Placebo (N=403)
Vestibular migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 5 mg (N=388) | Zavegepant 10 mg (N=394) | Zavegepant 20 mg (N=403) | Placebo (N=403)
Dysgeusia (Nervous system disorders) | 54 | 53 | 65 | 14
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 21 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03872453/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03872453/SAP_001.pdf